CLINICAL TRIAL: NCT00561886
Title: Change of Inspiratory Peak Flow After Bronchial Dilatation on Patients With Moderate to Severe COPD
Brief Title: Change of Inspiratory Peak Flow in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPF0601T; IPF0601T
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; lung function; dysnpea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients with COPD receiving once 24 µg formoterol
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Formoterol — One inhalation of 24µg Formoterol

SUMMARY:
Chronic obstructive bronchitis and emphysema (COPD) are pathophysiologically characterized by inflammatory and structural changes in the lung. These changes lead to a reduction in elastic recoil as well as reduction in lung parenchyma. As a consequence collapse of the small airway occurs during expiration leading to expiratory flow limitation. In severe cases this flow limitation occurs even during resting condition. This expiratory collapse is suspected to mask changes in bronchial smooth muscle tone, especially if these changes in bronchial smooth muscle tone are assessed using expiratory manoeuvres. This might leave the impression of non-reversible airway obstruction und ineffectiveness of treatment with bronchodilators. Several studies suggest that in patients with COPD symptomatic changes following application of a bronchodilating compound do not correlate with changes in forced expiratory volumes. In contrast inspiratory lung function parameters (especially forced inspiratory volume in one second (FIV1)) is much more associated with symptomatic changes in patients with COPD. Comparable effects were also detected regarding peak inspiratory flow (PIF) values.Changes in inspiratory parameters following administration of a bronchodilator in patients with COPD and asthma are reproducible. PIF can easily be measured by inspiratory peak flow meters. So far no data exists on the usability of these devices following bronchodilation in patients with COPD. Formoterol is a rapid acting bronchodilator, which has been proven save in asthma and COPD

DETAILED DESCRIPTION:
N=40 patients with moderate to severe COPD (30 < FEV1 < 70 % pred.), no further significant lung disease; current smokers or ex-smokers; no exacerbation in the last 2 month.

Baseline visit Physical examination Dsypnea score (Borg-Scale, TDI) Lung function (Bodyplethysmography, CO-diffusion capacity)

Before each study day the following medication will be withheld:

Short-acting bronchodilators > 6 hours Long-acting b2-adrenoceptor agonist > 24 hours Tiotropium > 24 hours

Study day 1 Bodyplethysmography including FEV1, PEF, FIV1 and PIF and assessment of PIF using an inspiratory Peak Flow Meter in randomized order.

Dysnpea Scores 30 minute break Assessment of change in dyspnea (visual analogue scale) Bodyplethysmography including FEV1, PEF, FIV1 and PIF. Assessment of PIF using an inspiratory Peak Flow Meter in randomized order Administration of 12 µg formoterol 30 minute break Assessment of change in dyspnea (visual analogue scale) Bodyplethysmography including FEV1, PEF, FIV1 and PIF. Assessment of PIF using an inspiratory Peak Flow Meter in randomized order.

Study day 2 Three to 14 days following study day 1. Schedule like day 1 with change in the order of lung function testing depending on randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with COPD of moderate to severe degree according to GOLD guidelines
2. current or ex-smokers, no history of atopy, stable clinical condition, age of >40 years.

Exclusion Criteria:

1. Significant lung disease other than COPD, unstable clinical condition
2. acute exacerbation in the last 2 month

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory peak flow following administration of a bronchodilator assessed by inspiratory peak flow device in patients with moderate to sever COPD | October 2007

SECONDARY OUTCOMES:
Correlation of changes in FEV1, FIV1 and PIF following bronchodilation in spirometry | October 2007
Correlation of change in PIF and symptomatic improvement in patients with COPD following bronchodilatation | October 2007

CONTACTS AND LOCATIONS:
Overall Officials: Roland Buhl, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Johannes Gutenberg-Univeristy, Mainz, Germany

REFERENCES:
- [Background] Taube C, Lehnigk B, Paasch K, Kirsten DK, Jorres RA, Magnussen H. Factor analysis of changes in dyspnea and lung function parameters after bronchodilation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 Jul;162(1):216-20. doi: 10.1164/ajrccm.162.1.9909054. PMID 10903244
- [Derived] Taube C, Rydzy L, Eich A, Korn S, Kornmann O, Sebastian M, Jorres RA, Buhl R. Use of a portable device to record maximum inspiratory flow in relation to dyspnoea in patients with COPD. Respir Med. 2011 Feb;105(2):316-21. doi: 10.1016/j.rmed.2010.11.017. Epub 2010 Dec 9. PMID 21145720